CLINICAL TRIAL: NCT01202396
Title: The Interaction Between the Intestinal Microbiota, Innate Defense and Epithelial Integrity in the Development of Pouchitis: a Multifactorial Approach
Brief Title: The Interaction Between Intestinal Microbiota, Innate Defense and Epithelial Integrity in the Development of Pouchitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. Dr. A. Masclee, Maastricht University Medical Center
Other Study IDs: MEC-10-2-033
Record Dates: First submitted 2010-09-02; First posted 2010-09-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Pouchitis
Keywords: pouch; pouchitis; ulcerative colitis; microbiota; defensins; epithelial integrity
MeSH Terms: conditions — Pouchitis; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In the prospective study the following biospecimens will be collected: faeces, serum, plasma, leucocytes, urine, intestinal biopsies and mucus

GROUPS / COHORTS (1):
- ulcerative colitis patients with a pouch: * ulcerative colitis patients undergoing proctocolectomy with an ileal pouch anal anastomosis
  * comparing patients with versus those without pouchitis
  * no intervention

SUMMARY:
Pouchitis is a common complication following proctocolectomy with ileal pouch anal anastomosis (IPAA) in patients with ulcerative colitis (UC). It affects the quality of life and can become a chronic problem. The aetiology of pouchitis is not completely understood. A crucial role of the intestinal microbiota has been suggested, but no causative agent has been identified so far. Furthermore, the defensin expression and the epithelial integrity are altered in inflammatory bowel diseases and may play an important role in the development of intestinal inflammation. Therefore, it has been hypothesized that the interaction between an altered microbiota composition, a defective epithelial integrity and changes in innate defense parameters such as defensins has a pivotal role in the development of pouchitis in UC patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with ulcerative colitis undergoing a total colectomy with IPAA for steroid dependent disease, therapy-refractory disease, colorectal cancer or severe dysplasia
* 18-65 years of age

Exclusion Criteria:

* unable to give informed consent
* pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing proctocolectomy with the construction of an ileal pouch anal anastomosis will be asked to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Differences in the intestinal microbiota composition between pouch patients with and without pouchitis | 24 months.
  A phylogenetic microarray will be used to characterize the luminal and mucosal microbiota composition (based on the SSU rRNA gene)of pouch patients with and without pouchitis. Anticipated results are the identification of specific bacterial profiles, genera and/or species dat are discriminating between subgroups.

SECONDARY OUTCOMES:
The expression of defensins in the intestinal mucosa | 24 months
  The mRNA expression levels of human alfa and beta-defensins in intestinal mucosal biopsies will be assessed by real time PCR
The intestinal permeability | 24 months.
  The epithelial integrity will be studied by the multiple sugar test to assess small intestinal and whole gut permeability.
Inflammatory mediators | 24 months
  Cytokine levels will be studied in serum and in intestinal biopsies. Furthermore, a histological evaluation and the MPO activity will be studied in these biopsies and calprotectin levels will be determined in 'fecal' sampels.
The expression of tight-junction associated proteins | 24 months.
  The intestinal tight junctions-associated proteins will be studied by immune staining of intestinal biopsies and mRNA levels in intestinal biopsies using real time PCR. Biopsies will be collected from standardised locations.

CONTACTS AND LOCATIONS:
Overall Officials: A. Masclee, Prof MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, div. Gastroenterology-Hepatology, Maastricht, Limburg, Netherlands